CLINICAL TRIAL: NCT07202338
Title: Is the Quality of the Therapeutic Alliance Associated With the Response to ChronoS Therapy? A Study in Patients With Mood Disorders
Brief Title: Association Between the Quality of the Therapeutic Alliance and the Response to ChronoS Therapy
Acronym: PREDI-CHRONOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D22_EPI0028_B
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Insomnia Related to Another Mental Condition
Keywords: Insomnia; Mood disorders; therapeutic alliance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Before/after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHRONOS therapy (Experimental)
  Interventions: Behavioral: CHRONOS therapy

INTERVENTIONS:
Behavioral: CHRONOS therapy — Description: Session 1 : Introduction and awareness of the sleep-wake link Session 2 : Awareness of day/night habits and behaviors Session 3 : Awareness of sleep/wake rhythms and sleepiness signals Session 4 : Awareness of the night/bed/sleep association Session 5 : Awareness of emotions and thoughts related to sleep Session 6 : Awareness of possible alternatives Session 7 : Awareness of one's relationship to sleep Session 8 : Awareness of future benefits

SUMMARY:
PREDI-CHRONOS is an ancillary study of the CHRONOS project (NCT07180290) The goal of this study is to measure the association between therapeutic alliance and the clinical response to the CHRONOS therapy.

The CHRONOS therapy is a new psychotherapy integrating:

1. Interpersonal and Social Rhythm Therapy
2. Chronotherapies to regulate sleep/wake cycles
3. Positive mental imagery for stress management
4. Mindfulness therapy for both stress and hyperarousal state management This therapy applied to patients with mood disorders (uni- or bipolar disorder). All participants in the study underwent the therapy. Response was defined as an improvement in the Insomnia Severity Index (ISI) from baseline to the end of the study.

The aim is to study the association of the therapeutic alliance with the response to the CHRONOS therapy, using the working alliance inventory (WAI) questionnaire.

Secondary objectives were to identify other factors potentially associated with the response to the therapy: history of a trauma, emotional regulation, and time perspective.

DETAILED DESCRIPTION:
Insomnia affects 85% of patients with a mood disorder during depressive phases and more than 50% will suffer from insomnia symptoms after remission. The treatment of insomnia with mood disorders represents a major therapeutic issue. European recommendations suggest that cognitive behavioural therapy for insomnia (iCBT) as the first-line reference treatment for chronic insomnia disorder. However, only 38% of patients respond positively to the treatment at 24 months, while 50% of patients with insomnia disorder and mood disorder do not respond to the treatment.

A new psychotherapy was developed within the Psychiatry, Sleep and Chronobiology Reference Center (ChronoS) integrating:

1. Interpersonal and Social Rhythm Therapy
2. Chronotherapies to regulate sleep/wake cycles
3. Positive mental imagery for stress management
4. Mindfulness therapy for both stress and hyperarousal state management The investigators designed a "before/after" study to evaluate the effectiveness of this psychotherapy with multimodal approaches on the severity of insomnia in patients with mood disorders (CHRONOS study, NCT07180290).

PREDI-CHRONOS is an ancillary study aiming at evaluating the association between therapeutic alliance and the clinical response to the CHRONOS therapy. Therapeutic alliance (or working alliance) can be defined as the collaborative relationship between patient and therapist based on purposeful collaboration and an affective bond. It is known to play an important role in therapeutic progress and treatment success.

Population: PREDI-CHRONOS included all patients that underwent the CHRONOS therapy (patients >= 18 years old, with mood disorders and an Insomnia Index Score >= 8, indicating the presence of insomnia). Patients under protection measures (curatorship) were not included in the study.

Main objective: to measure the correlation between the therapeutic alliance and the response to the CHRONOS therapy. Response was defined as an improvement in the Insomnia Severity Index (ISI) from baseline to the end of the study. Therapeutic alliance was measured using the Working Alliance Inventory (WAI) questionnaire.

Secondary objectives: to identify other factors potentially associated with the response to the therapy: history of a trauma, emotional regulation, and time perspective.

PREDI-CHRONOS design is similar as CHRONOS study, a first visit (V0) was scheduled before the start of the CHRONOS therapy (pre-intervention measures), then two visits at the beginning (V1) and the end (V2) of the therapy, and a final one 3 months after the end of the therapy (post-intervention measures).

Some data collected for CHRONOS study were used to characterise patients on other factors (anxiety and depressive symptoms, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with mood disorders diagnosed according to DSM-5 criteria
* Patients with insomnia based on a ISI score >= 8

Exclusion Criteria:

* Patients < 18 years old
* Patients with psychotic disorders
* Patients who have previously received cognitive therapy for insomnia
* Patient subject to protective measures (curatorship)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Response to CHRONOS therapy | Visit 1 : 1st session of the CHRONOS therapy (4 to 6 weeks after inclusion) Visit 2 : last session of the CHRONOS therapy (8 weeks after V1)
  Response to therapy was measured by the Insomnia Severity Index (ISI). The score ranging from 17 to 84. A score above 7 indicating the presence of insomnia (score between 8-14 = insomnia symptoms of mild to moderate severity; score between 15-21 = insomnia symptoms of moderate severity; score between 22-28 = severe insomnia symptoms) An improvement in the ISI score between the beginning and the end of the therapy was considered as an effective response
Evaulation of therapeutic alliance | Visit 1: 1st session of the CHRONOS therapy (4 to 6 weeks after inclusion) Visit 2: last session of the CHRONOS therapy (8 weeks after V1)
  Therapeutic alliance was measured using the Working Alliance Inventory Short Revised (WAI-SR), a 12-item form, and scores ranging from 5 to 20. Higher scores indicate a better therapeutic alliance.

SECONDARY OUTCOMES:
Presence of a trauma | Visit 1 : 1st session of CHRONOS therapy (4 to 6 weeks after inclusion)
  The Adversed Childhood Experiences (ACE) questionnaire is a 10-item self-report tool, which is a count of the total number of adverse events respondents reported.
Emotional regulation | Visit 1 : 1st session of CHRONOS therapy (4 to 6 weeks after inclusion) Visit 2 : last session of CHRONOS therapy (8 weeks after V1)
  Questionnaires Difficulties in Emotion Regulation Scale (DERS). A total score is calculated by summing the item responses and ranges from 18 to 90; higher scores indicate greater difficulty with emotion regulation.
Time perspective | Visit 1: 1st session of CHRONOS therapy (4 to 6 weeks after inclusion)
  Zimbardo Time Perspective Inventory (ZTPI). The questionnaire distinguished five time perspectives (past-negative, past-positive, present-hedonistic, present-fatalistic, and future). Well-being was reflected by a balanced time perspective (BTP). Deviation from the balanced time perspective is defined as a Euclidean distance between optimal (o) and empirical (e) levels of time perspectives.
  Results showed that balanced time perspective is associated with greater past positive (PP) and future (F) and lower past negative (PN) and present fatalistic (PF) time perspectives.
Presence of a trauma | Visit 1: 1st session of the CHRONOS therapy (4 to 6 weeks after inclusion)
  PTSD Checklist for DSM-5 (PCL-5): Several criteria (exposition to a traumatic vent, re-experienced traumatic event, negative thoughts, etc.) allow to identify posttraumatic stress disorder among adults. All of the criteria are required for the diagnosis of PTSD.
Emotional regulation | Visit 1 : 1st session of CHRONOS therapy (4 to 6 weeks after inclusion) Visit 2 : last session of CHRONOS therapy (8 weeks after V1)
  Emotion regulation questionnaire (ERQ). Respondents' answers are scored on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scoring takes the average of all the scores in each subscale. A higher score indicate greater use of emotion regulation strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Paris Psychiatrie et Neurosciences, Paris, France

IPD SHARING:
Plan to Share IPD: No